CLINICAL TRIAL: NCT03484455
Title: A Prospective Randomized Multi-Center Study of the Use of the Organ Recovery Systems LifePort® Liver Transporter (LLT) System With Vasosol® as Compared to Static Cold Storage in Orthotopic Liver Transplants (Perfusion to Improve Liver Outcomes in Transplantation)
Brief Title: Study to Evaluate Performance of the Organ Recovery Systems LifePort® Liver Transporter System, a Machine Perfusion System, for Liver Transplant
Acronym: PILOT™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organ Recovery Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-US-01-ORS
Record Dates: First submitted 2018-03-02; First posted 2018-03-30 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Hypothermic Machine Perfusion (Experimental): Hypothermic Machine Perfusion with Organ Recovery Systems LLT system
  Interventions: Device: Hypothermic machine perfusion
- Static Cold Storage (Active Comparator): Standard of Care - Static Cold Storage
  Interventions: Device: Static cold storage

INTERVENTIONS:
Device: Hypothermic machine perfusion — Organ Recovery Systems LifePort® Liver Transporter (LLT) System and Vasosol® Machine Perfusion Solution
  Arms: Hypothermic Machine Perfusion
Device: Static cold storage — Static cold storage (standard of care)
  Arms: Static Cold Storage

SUMMARY:
Comparison of hypothermic machine perfusion of livers to standard of care (static cold storage).

DETAILED DESCRIPTION:
Prospective, randomized, multi-center study to show safe and effective use of whole liver preservation via hypothermic machine perfusion (HMP) as compared to livers preserved by static cold storage.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Active on the United Network for Organ Sharing (UNOS) waiting list for liver transplantation
* De novo liver transplant recipient
* Written informed consent required

Exclusion Criteria:

* Subject is a multi-organ transplant recipient
* Subject is antibodies blood group (ABO) liver incompatible
* Subject has severe systemic infection
* Subject is Human Immunodeficiency Virus (HIV) positive
* Subject has acute/fulminant liver failure
* Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Number of patients in each arm with Early Allograft Dysfunction (EAD) | 7 days
  EAD defined as total bilirubin ≥ 10 mg/dL or International Normalized Ratio (INR) ≥ 1.6 or Aspartate Aminotransferase (AST) >2000IU/L or Alanine Aminotransferase (ALT) > 2000 IU/L

CONTACTS AND LOCATIONS:
Overall Officials: Stan Harris, Study Director — Organ Recovery Systems; Matthew Copithorne, Study Chair — Organ Recovery Systems
Locations (9):
- United States (9):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - University of Rochester Strong Memorial Hospital, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia Hospital, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No